CLINICAL TRIAL: NCT06936969
Title: Comparison of 40% Glucose Solution and Autologous Blood Patch Pleurodesis for Postoperative Air Leak After Lung Resections: Prospective Randomized Study
Brief Title: Comparison of 40% Glucose Solution and Autologous Blood Patch Pleurodesis for Postoperative Air Leak After Lung Resections
Acronym: GLUC-PAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wielkopolskie Centrum Pulmonologii i Torakochirurgii (Other)
Collaborators: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 765/24
Record Dates: First submitted 2025-03-28; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: Prolonged Air Leak; Persistent Air Leak
Keywords: PAL; ABPP; Prolonged air leak; persistent air leak; lung cancer; anatomical lung resection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: patients with PAL in whom pleurodesis was performed using autologous blood (ABPP). (Active Comparator): After obtaining informed consent, the patient will lie supine in their room. 30 minutes before the procedure, the patient's capillary blood glucose level will be measured. The patient does not have to fast before the procedure. The nurse will be asked to collect 120 ml of peripheral venous blood from the patient. Then the doctor, assisted by the nurse, will first administer 20 ml of 1% Lignocaine through the pleural drain, and then after about 5-10 minutes, the patient's previously collected venous blood. At the moment of blood administration, the drainage system will be disconnected. Then, the drain will be "injected" with 20 ml of air to avoid clogging the drain. The patient will remain supine for two hours post-procedure, maintaining fasting status. After 30 minutes from the administration of the patient's own blood, the capillary blood glucose level will be measured again. After two hours, the patient, with nursing assistance, may resume normal activities.
  Interventions: Procedure: Autologous blood patch pleurodesis
- Study group: Patients in whom pleurodesis was performed using a 40% glucose solution. (Experimental): After obtaining informed consent, the patient will lie supine in their room. Thirty minutes prior to the procedure, a capillary blood glucose measurement will be taken; fasting is unnecessary. Initially, 20 ml of 1% lignocaine will be administered via the pleural drain. After a 5-10 minute interval, 120 ml of a 40% glucose solution (Glucose 40 B. Braun 400 mg/ml for infusion, Ecoflac Plus) will be infused using two separate Luer Lock syringes to prevent cross-contamination. At the time of glucose administration, the drainage system will be temporarily disconnected. Subsequently, 20 ml of air will be introduced into the drain to prevent occlusion. The patient will remain supine and refrain from sitting or rotating for two hours post-procedure, maintaining fasting status. Capillary blood glucose will be re-assessed 30 minutes after glucose administration. After two hours, the patient, with nursing assistance, may resume normal activities.
  Interventions: Procedure: 40% glucose solution pleurodesis

INTERVENTIONS:
Procedure: Autologous blood patch pleurodesis — The intervention in this study is distinguished by the fact that patients are randomized, the dose of both glucose and ABPP is 120 ml, the patient remains in a supine position for 2 hours after administration, the procedure can be repeated at 48-hour intervals, a maximum of 3 times.
  Other Names: ABPP; bloodpatch
  Arms: Control group: patients with PAL in whom pleurodesis was performed using autologous blood (ABPP).
Procedure: 40% glucose solution pleurodesis — After obtaining informed consent, the patient will lie supine in their room. 30 minutes before the procedure, the patient's capillary blood glucose level will be measured. The patient does not have to fast before the procedure. The nurse will be asked to collect 120 ml of peripheral venous blood from the patient. Then the doctor, assisted by the nurse, will first administer 20 ml of 1% Lignocaine through the pleural drain, and then after about 5-10 minutes, the patient's previously collected venous blood. At the moment of blood administration, the drainage system will be disconnected. Then, the drain will be "injected" with 20 ml of air to avoid clogging the drain. The patient will remain supine for two hours post-procedure, maintaining fasting status. After 30 minutes from the administration of the patient's own blood, the capillary blood glucose level will be measured again. After two hours, the patient, with nursing assistance, may resume normal activities.
  Other Names: chemical pleurodesis; glucose solution pleurodesis
  Arms: Study group: Patients in whom pleurodesis was performed using a 40% glucose solution.

SUMMARY:
Prolonged or persistent air leak (PAL) is one of the most common complications in patients after surgery on the lung parenchyma. Air leaks typically originate from alveolar-pleural fistulas, which can result from surgical manipulation of the lung parenchyma or the bronchial stump after procedures such as lobectomy. Key risk factors for PAL include extensive lung resections such as lobectomy, presence of pleural adhesions, incomplete interlobar fissures, chronic obstructive pulmonary disease (COPD), asthma, emphysema, advanced age, and reduced preoperative lung function, particularly low preoperative FEV1 values.

PAL necessitates extended pleural drainage, leading to significant patient discomfort, pain, and substantial limitations in early postoperative rehabilitation. In patients with pre-existing pulmonary conditions like bronchial asthma or COPD, PAL can markedly worsen clinical status, resulting in severe complications such as infections, pneumonia, pleural empyema, acute respiratory distress syndrome, and even mortality. In extreme cases, PAL may contraindicate chemotherapy, causing significant delays in adjuvant therapy post-surgery. Effective management of PAL can significantly enhance patient quality of life, facilitating a quicker return to normal activities and continuation of systemic treatment.

Moreover, PAL is a leading cause of extended hospitalization, invariably increasing treatment costs. Therefore, the necessity for safe and effective treatment of PAL is justified not only medically but also economically.

Current standards for PAL treatment encompass both surgical and non-surgical methods. The available literature describes various conservative treatments, among which pleurodesis is commonly employed. Non-surgical pleurodesis techniques include the intrapleural administration of the patient's autologous blood or chemical agents such as medical talc, povidone-iodine, or doxycycline.

Intrapleural administration of autologous blood, known as autologous blood patch pleurodesis (ABPP), is widely utilized for the conservative treatment of PAL. This method involves injecting the patient's own blood into the pleural space through an existing chest tube, promoting clot formation and sealing of the air leak. Studies have demonstrated the safety and efficacy of ABPP, with success rates exceeding 80% in sealing air leaks within 48 hours and a low incidence of complications such as fever or empyema.

Another method highlighted in limited scientific literature is the intrapleural administration of a 50% glucose solution. This technique has been primarily reported by authors from Asian countries, such as Japan and Korea, and is not widely adopted in Western centers. Available studies emphasize its effectiveness, with success rates exceeding 80%, and report a lack of complications in patients undergoing pleurodesis with concentrated glucose solutions.

The aim of our study is to compare the effectiveness of a 40% glucose solution with the ABPP. The selection of a 40% glucose solution is due to the unavailability of a 50% glucose solution in the Polish pharmaceutical market.

Potential benefits of effective PAL treatment include improved patient quality of life, reduced hospitalization duration, decreased risk of complications, and lower treatment costs. Prolonged hospitalization and treatment associated with PAL generate significant expenses for the healthcare system. Our study may contribute to significant improvements in treatment outcomes, patient quality of life, and the cost-effectiveness of thoracic surgical procedures. In the long term, this research may also influence the development of new treatment standards and clinical protocols.

DETAILED DESCRIPTION:
Prolonged or persistent air leak (PAL) is one of the most common complications in patients after surgery on the lung parenchyma. Air leaks typically originate from alveolar-pleural fistulas, which can result from surgical manipulation of the lung parenchyma or the bronchial stump after procedures such as lobectomy. PAL incidence ranges from 5% to 25% of all pulmonary resection procedures. The air leak typically originates from alveolar-pleural fistulas, representing a communication between distal pulmonary alveoli and the pleural space, often occurring along the mechanical suture line or its vicinity.

Prolonged or persistent air leak (PAL) is one of the most common complications in patients after lung parenchyma surgery. PAL is defined as the loss of air from the residual lung parenchyma, persisting beyond the fifth day after surgery. PAL incidence ranges from 5% to 25% of all pulmonary resection procedures. The source of the air leak may be the lung parenchyma damaged as a result of surgical manipulation or the stump of the severed bronchus. In most cases, The air leak typically originates from alveolar-pleural fistulas, representing a communication between distal pulmonary alveoli and the pleural space, often occurring along the mechanical suture line.

Key risk factors for PAL include extensive pulmonary resections (e.g., lobectomy), presence of pleural adhesions, incomplete interlobar fissures, chronic obstructive pulmonary disease (COPD), asthma, pulmonary emphysema, advanced age, and reduced preoperative pulmonary function, particularly low preoperative FEV1 values.

PAL necessitates prolonged pleural drainage, leading to patient discomfort, pain, and significant limitations in early postoperative rehabilitation. In patients with pre-existing pulmonary conditions (e.g., asthma, COPD), PAL can severely deteriorate clinical status, potentially causing infections, pneumonia, pleural empyema, acute respiratory distress syndrome, or even death. Additionally, prolonged air leaks may contraindicate chemotherapy and delay adjuvant therapy post-surgery. Effective PAL management can enhance patient quality of life, facilitate quicker recovery, and allow timely continuation of systemic treatments.

PAL is a leading cause of extended hospital stays, increasing healthcare costs. Therefore, safe and effective PAL management is justified both medically and economically.

Current PAL treatment standards include surgical and non-surgical methods. Intraoperative techniques to prevent air leaks encompass pleural tenting (especially during upper lobectomies), reinforcement or suturing of stapler lines, fissure-less techniques, and the use of tissue adhesives or specialized aerostatic dressings. Some patients with PAL may require reoperation, involving the aforementioned methods or direct suturing of the air leak site using manual or mechanical staplers. However, reoperations after pulmonary parenchymal resections often present more challenging conditions than the initial surgery and may introduce additional complications and psychological stress for the patient.

Notably, air leaks from alveolar-pleural fistulas may go undetected during surgery, and preventive strategies cannot always be applied intraoperatively. Consequently, much of the available literature focuses on conservative postoperative PAL management. Non-surgical methods, such as pleurodesis, involve intrapleural administration of agents like autologous blood, medical talc, povidone-iodine, or doxycycline.

Talc pleurodesis is a preferred method in many centers for treating spontaneous pneumothorax and recurrent pleural effusions. Studies have reported its efficacy in PAL treatment, with success rates exceeding 90%. However, concerns exist regarding potential long-term side effects due to systemic talc distribution and accumulation in organs such as the liver, kidneys, spleen, bone marrow, or brain. While animal studies have highlighted these risks, similar human studies are lacking, and there is insufficient evidence confirming talc's harm in these locations. Nonetheless, the absence of long-term follow-up studies on medical talc administration warrants caution, especially in younger patients with extended life expectancy.

A less invasive approach is pleurodesis using intrapleural administration of the patient's autologous blood (ABPP). This globally practiced conservative PAL treatment lacks high-quality randomized studies and large-scale longitudinal research. Nevertheless, it is often perceived as safe within the thoracic surgery community, with most studies highlighting its high efficacy. Advantages include bedside administration, repeatability every 48 hours, no risk of anaphylaxis, and a generally low complication rate, although potential side effects include fever, pleural effusion, or pleural empyema.

Another method demonstrating efficacy and safety in limited studies is intrapleural administration of a 50% glucose solution. Predominantly utilized by authors from Asian countries (Japan, Korea), this technique appears underreported in Western centers, as evidenced by the lack of related studies from these regions. Available research indicates an efficacy rate exceeding 80% and an absence of complications following pleurodesis with concentrated glucose solution. A comparative study by Hong et al. involving 100 patients (64 receiving autologous blood pleurodesis and 36 receiving 50% glucose solution pleurodesis) reported comparable efficacy and safety between the two methods. However, a 1992 case from China documented acute pneumonia following 50% glucose administration to treat an air leak during a first episode of pneumothorax. Due to the irritant properties of the glucose solution, authors emphasize the necessity of prior anesthesia using intrapleural administration of 20 ml of 1% lignocaine to alleviate potential pain.

Our study aims to compare the efficacy of a 40% glucose solution with the ABPP. The choice of a 40% glucose solution is dictated by the unavailability of a 50% glucose solution in the Polish pharmaceutical market.

Effective PAL treatment offers potential benefits, including improved patient quality of life, reduced hospitalization duration, decreased complication risks, and lower treatment costs. Research into air leaks, a frequent and costly complication leading to numerous medical issues, is crucial. Studies on PAL contribute to a better understanding of the physiological and pathological mechanisms associated with postoperative wound healing within the thoracic cavity, particularly the pulmonary parenchyma. Research should not only assess method efficacy but also identify factors influencing pleurodesis success, such as surgical techniques, comorbidities, and timing of the pleurodesis-inducing agent administration.

Prolonged hospitalization and treatment due to PAL generate significant healthcare costs. Establishing a standard treatment method that is safe, effective, affordable, and readily available could substantially improve the treatment process for oncology patients, reduce hospital stay costs, and decrease the need for additional medical procedures. Investigating new PAL treatment methods after thoracic surgeries is vital from clinical, scientific, and economic perspectives. Potential benefits from our study may include significant improvements in treatment outcomes, patient quality of life, and cost-effectiveness of thoracic surgery procedures. In the long term, this research could also influence the development of new treatment standards and clinical protocols.

ELIGIBILITY:
Inclusion Criteria:

* Age: patients aged 18 years or older.
* Surgical Procedure: patients who underwent anatomical lung resections (segmentectomy, lobectomy, or bilobectomy) at the Department of Thoracic Surgery, Poznan University of Medical Sciences, between November 2023 and December 2024.
* Prolonged Air Leak Diagnosis: patients with diagnosed PAL after lung resection, as defined by air leakage persisting beyond 5 days post-surgery.
* Consent: patients who were willing to provide informed consent for participation in the study and for the intervention procedures (autologous blood pleurodesis or 40% glucose solution pleurodesis).

Exclusion Criteria:

* Non-Anatomical Resections: Patients who underwent non-anatomical resections, such as pneumonectomy, lung transplantation, sleeve resections, or wedge resections.
* Patients from whom the required volume of peripheral blood (120 ml) could not be collected.
* Active Infection or Sepsis: Patients with ongoing infections or sepsis at the time of enrollment.
* Reoperation or Additional Interventions: patients who required immediate reoperation or other interventions that disturb the process of treating PAL.
* Mental Health or Cognitive Impairment: patients with significant cognitive impairments or mental health conditions that hinder the ability to provide informed consent or comply with study procedures.
* Patients who failed to perform three ABPP or 40% glucose injections (no consent, need for urgent surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of Days Until Resolution of Prolonged Air Leak (PAL) | From date of randomization up to 90 days from the procedure
  The primary endpoint is the resolution of postoperative air leak after a maximum of three administrations of autologous blood pleurodesis (ABPP) or a 40% glucose solution. Resolution is defined as an air leak rate of less than 20 mL/min for at least 8 hours, successful drain removal, no pneumothorax on a control X-ray taken 3 hours after drain removal, and the patient's discharge home.

SECONDARY OUTCOMES:
Incidence of complications, number of days of prolonged chest drainage and length of inhospital stay (in days). | From the date of randomization until 90 days following the procedure.
  pain intensity, complications related to the administration of autologous blood or 40% glucose solution, postoperative complications (such as residual pleural space persistence, need for repeated pleural drainage), drainage duration, hospitalization length, and the absence of re-drainage or additional surgical intervention. This included reoperation within 90 days of surgery due to persistent residual pleural space or the occurrence of pneumothorax.

CONTACTS AND LOCATIONS:
Locations (1):
- Wielkopolskie Centrum Pulmonologii i Torakochirurgii, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skrzypczak PJ, Dobiecki T, Rozmiarek M, Gabryel P, Kasprzyk M, Piwkowski C. Comparison of 40% Glucose Solution and Autologous Blood Patch Pleurodesis for the Treatment of Postoperative Air Leak After Lung Resections: A Prospective Randomized Controlled Study. Eur J Cardiothorac Surg. 2025 Nov 2;67(11):ezaf382. doi: 10.1093/ejcts/ezaf382. PMID 41191623